CLINICAL TRIAL: NCT00453973
Title: An Open-Label, Multi-Center, Extension Study to Evaluate the Safety and Tolerability of Peginesatide for the Long-Term Maintenance Treatment of Anemia in Patients With Chronic Kidney Disease
Brief Title: Extension Study to Evaluate Safety and Tolerability of Peginesatide for Long-Term Treatment of Anemia in Participants With CKD (EU)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to more robust long-term data generated in other active-controlled studies
Sponsor: Affymax (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFX01-10; 2006-003846-41 (EudraCT Number)
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Renal Failure; Chronic Kidney Disease; Anemia
Keywords: anemia; chronic kidney disease; CKD; chronic renal failure; CRF; dialysis; erythropoietin; EPO; erythropoiesis stimulating agent; ESA; Hematide™; hemodialysis; hemoglobin; Hb; Hgb; Omontys; peginesatide; red blood cell; red blood cell production
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Anemia | interventions — peginesatide; hematide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maintenance Switch in Dialysis Participants (Experimental): Participants were from a prior Affymax peginesatide treatment study conducted in participants who were on dialysis and had been on Epoetin at study entry, and who were switched to peginesatide (NCT00434330). This group is categorized as "Maintenance Switch in Dialysis Participants" regardless of dialysis status at the start of or during this study.
  Interventions: Drug: peginesatide
- Treatment Initiation in Non-Dialysis Participants (Experimental): Participants were from a prior Affymax peginesatide treatment study conducted in participants who were not on dialysis and not on erythropoiesis stimulating agents (ESAs), and who received peginesatide (NCT00228436). This group is categorized as "Initiation of Treatment in Non-Dialysis Participants" regardless of dialysis status at the start of or during this study.
  Interventions: Drug: peginesatide

INTERVENTIONS:
Drug: peginesatide — Participants received the same initial peginesatide dose via the same route, intravenously or subcutaneously, as was administered at the end of the previous peginesatide treatment study in which the participant was enrolled. The median first dose at study start was 0.044 milligram per kilogram (mg/kg) with an interquartile range of 0.028 to 0.076 mg/kg. Each participant was to receive peginesatide as an injection administered once every 4 weeks for approximately 54 months in this trial.
  Other Names: Omontys; Hematide; AF37702 Injection
  Arms: Maintenance Switch in Dialysis Participants
Drug: peginesatide — Participants received the same initial peginesatide dose via the same route, intravenously or subcutaneously, as was administered at the end of the previous peginesatide treatment study in which the participant was enrolled. The median first dose at study start was 0.024 mg/kg with an interquartile range of 0.017 to 0.035 mg/kg. Each participant was to receive peginesatide as an injection administered once every 4 weeks for approximately 54 months in this trial.
  Other Names: Omontys; Hematide; AF37702 Injection
  Arms: Treatment Initiation in Non-Dialysis Participants

SUMMARY:
The purpose of this study was to evaluate the long term safety and tolerability of peginesatide for the maintenance of hemoglobin in participants with chronic kidney disease (CKD) who had received at least 24 weeks of peginesatide treatment in an earlier study.

DETAILED DESCRIPTION:
Anemia associated with chronic kidney disease is due to several factors, primarily the inability of the diseased kidneys to produce adequate amounts of endogenous erythropoietin. Ancillary factors include the shortened lifespan of red blood cells, iron and other nutritional deficiencies, infection, and inflammation. The presence and severity of anemia are related to the duration and extent of kidney failure. Anemia is associated with increased mortality, increased likelihood of hospitalization, reduced cognitive function, and increased left ventricular hypertrophy and heart failure.

Erythropoiesis stimulating agents (ESAs) have been established as a treatment for anemia in subjects with chronic kidney disease, and have improved the management of anemia over alternatives such as transfusion. Peginesatide is a parenteral formulation developed for the treatment of anemia associated with chronic kidney disease. Peginesatide binds to and activates the human erythropoietin receptor, and stimulates erythropoiesis in human red cell precursors in a manner similar to other known erythropoiesis-stimulating agents.

Study participants had received at least 24 weeks of peginesatide dosing in a previous Affymax-sponsored study and were to receive doses of peginesatide for up to 54 months. However, the Sponsor ended the study early.

ELIGIBILITY:
Inclusion Criteria:

* Participant is informed of the investigational nature of this study and has given written, informed consent in accordance with institutional, local, and national guidelines.
* Males or females ≥ 18 years of age.
* Premenopausal females (with the exception of those who are surgically sterile) must have a negative pregnancy test at screening; those who are sexually active must practice a highly effective method of birth control for at least 4 weeks prior to study drug administration, and must be willing to continue contraception until at least 4 weeks after the last dose of study drug.
* Participant who has received at least 24 weeks of peginesatide dosing in a previous Affymax-sponsored study.
* One hemoglobin value of ≥ 10.0 grams per deciliter (g/dL) in the 4 weeks prior to study drug administration.

Exclusion Criteria:

* Known intolerance to peginesatide or pegylated products.
* History of antibodies to any erythropoiesis stimulating agent (ESA) or history of pure red cell aplasia (PRCA).
* High likelihood of early withdrawal or interruption of the study (e.g., participant suffers from any clinically significant medical disease or condition that may, in the Investigator's opinion, interfere with safety, assessment, or follow-up of the participant)
* Anticipated life expectancy < 18 months
* Receipt of any ESA other than peginesatide at any time after participant enrollment in the previous Affymax-sponsored study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2006-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President, Clinical Development, Study Director — Affymax
Locations (18):
- Bulgaria (6):
  - Research Facility, Burgas
  - Research Facility, Pleven
  - Research Facility, Plovdiv
  - Research Facility, Rousse
  - Research Facility, Varna
  - Research Facility, Veliko Tarnovo
- Poland (3):
  - Research Facility, Bialystok
  - Research Facility, Katowice
  - Research Facility, Lodz
- Romania (5):
  - Research Facility, Arad
  - Research Facility, Bacau
  - Research Facility, Bucharest
  - Research Facility, Iași
  - Research Facility, Timișoara
- United Kingdom (4):
  - Research Facility, Croydon
  - Research Facility, Derby
  - Research Facility, London
  - Research Facility, Swansea

RESULTS

PARTICIPANT FLOW:
Groups:
- Maintenance Switch in Dialysis Participants: Participants were from a prior Affymax peginesatide treatment study conducted in participants who were on dialysis and had been on Epoetin at study entry, and who were switched to peginesatide (NCT00434330). The median first dose at study start was 0.044 milligram per kilogram (mg/kg) with an interquartile range of 0.028 to 0.076 mg/kg. This group is categorized as "Maintenance Switch in Dialysis Participants" regardless of dialysis status at the start of or during this study.
- Treatment Initiation in Non-Dialysis Participants: Participants were from a prior Affymax peginesatide treatment study conducted in participants who were not on dialysis and not on erythropoiesis stimulating agents (ESAs), and who received peginesatide (NCT00228436). The median first dose at study start was 0.024 mg/kg with an interquartile range of 0.017 to 0.035 mg/kg. This group is categorized as "Initiation of Treatment in Non-Dialysis Participants" regardless of dialysis status at the start of or during this study.
Period: Overall Study
Arm/Group | Maintenance Switch in Dialysis Participants | Treatment Initiation in Non-Dialysis Participants
Started | 51 | 63
Completed | 0 | 15
Not Completed | 51 | 48
Not completed — Adverse Event | 4 | 9
Not completed — Withdrawal by Subject | 7 | 6
Not completed — PI Decision | 0 | 2
Not completed — Relocation | 1 | 0
Not completed — Renal transplant | 1 | 1
Not completed — Site closed by sponsor | 3 | 0
Not completed — Sponsor Decision to Terminate Study | 35 | 30

BASELINE CHARACTERISTICS:
Arm/Group | Maintenance Switch in Dialysis Participants | Treatment Initiation in Non-Dialysis Participants | Pooled AF37702 Inj.
Number analyzed (Participants) | 51 | 63 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 22 | 64
  >=65 years | 9 | 41 | 50
Age Continuous [Mean (Standard Deviation); unit: years] | 53.2 (11.92) | 66.4 (13.48) | 60.5 (14.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 34 | 53
  Male | 32 | 29 | 61

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Mean Hemoglobin in the Target Range of 10.0-12.0 Grams Per Deciliter (g/dL) After Final Dosing Guideline Change
Time Frame: Up to 54 months
Population: Full Analysis - Number of participants with hemoglobin assessed after dosing guideline change
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance Switch in Dialysis Participants | Treatment Initiation in Non-Dialysis Participants
Number analyzed (Participants) | 28 | 40
percentage of participants | 0.786 | 0.875

ADVERSE EVENTS:
Arm/Group | Maintenance Switch in Dialysis Participants | Treatment Initiation in Non-Dialysis Participants
Serious Adverse Events (participants affected / at risk) | 10/51 | 31/63
Other Adverse Events (participants affected / at risk) | 46/51 | 55/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maintenance Switch in Dialysis Participants (N=51) | Treatment Initiation in Non-Dialysis Participants (N=63)
Atrial fibrillation (Cardiac disorders) | 2 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Aortic valve disease (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Pericardial haemorrhage (Cardiac disorders) | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
Catheter related complication (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Arteriovenous fistula site infection (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Pyelonephritis chronic (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetic foot (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal ganglia haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 2
Azotaemia (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Maintenance Switch in Dialysis Participants (N=51) | Treatment Initiation in Non-Dialysis Participants (N=63)
Angina pectoris (Cardiac disorders) | 3 | 2
Vertigo (Ear and labyrinth disorders) | 4 | 1
Hyperparathyroidism secondary (Endocrine disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 10 | 10
Abdominal pain (Gastrointestinal disorders) | 9 | 3
Abdominal pain upper (Gastrointestinal disorders) | 6 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 4
Vomiting (Gastrointestinal disorders) | 5 | 5
Toothache (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 0 | 4
Chest pain (General disorders) | 5 | 1
Catheter site haemorrhage (General disorders) | 4 | 0
Influenza like illness (General disorders) | 2 | 4
Fatigue (General disorders) | 1 | 6
Oedema peripheral (General disorders) | 1 | 12
Bronchitis (Infections and infestations) | 9 | 7
Tracheobronchitis (Infections and infestations) | 6 | 0
Hepatitis C (Infections and infestations) | 5 | 0
Tooth abscess (Infections and infestations) | 5 | 0
Respiratory tract infection viral (Infections and infestations) | 4 | 0
Urinary tract infection (Infections and infestations) | 4 | 7
Catheter related infection (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 1 | 13
Influenza (Infections and infestations) | 0 | 9
Lower respiratory tract infection (Infections and infestations) | 0 | 5
Procedural hypertension (Injury, poisoning and procedural complications) | 9 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 7 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 6 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 6 | 2
Procedural hypotension (Injury, poisoning and procedural complications) | 4 | 1
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 3 | 0
Procedural headache (Injury, poisoning and procedural complications) | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 4
Fall (Injury, poisoning and procedural complications) | 0 | 4
Blood pressure increased (Investigations) | 6 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 4
Gout (Metabolism and nutrition disorders) | 0 | 5
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 22 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 5
Headache (Nervous system disorders) | 28 | 5
Dizziness (Nervous system disorders) | 3 | 5
Insomnia (Psychiatric disorders) | 4 | 3
Renal failure (Renal and urinary disorders) | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 11 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 6
Hypertensive crisis (Vascular disorders) | 19 | 0
Hypotension (Vascular disorders) | 19 | 4
Hypertension (Vascular disorders) | 4 | 13

LIMITATIONS AND CAVEATS:
Early termination of study due to generation of controlled long-term data in Phase 3 studies. Amended dosing guidelines during the trial to reflect label changes for ESAs; the primary outcome was assessed after the dosing guideline change.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications may not contain Sponsor confidential information, and will be subject to Sponsor review prior to submission for publication.